CLINICAL TRIAL: NCT01990079
Title: Use of Technological Advances to Prevent Smoking Relapse Among Smokers With PTSD
Acronym: QUIT4EVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048990
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: PTSD; Smoking
Keywords: PTSD; smoking
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Smoking | interventions — Bupropion; Nicotine Replacement Therapy; Nicotine Chewing Gum; Transdermal Patch; Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- QUIT4Ever (Experimental): QUIT4EVER is an intervention that combines 4 guideline-based smoking cessation counseling sessions, bupropion and nicotine replacement therapy, mobile contingency management, and the smart-phone application Stay Quit Coach.
  Interventions: Drug: Bupropion; Drug: nicotine replacement therapy; Other: Smoking cessation counseling; Behavioral: mobile contingency management; Other: Stay Quit Coach
- Control Contact Condition (Active Comparator): This intervention combines 4 guideline-based smoking cessation counseling sessions, bupropion and nicotine replacement therapy, and mobile contingency management.
  Interventions: Drug: Bupropion; Drug: nicotine replacement therapy; Other: Smoking cessation counseling; Behavioral: mobile contingency management

INTERVENTIONS:
Drug: Bupropion — All participants who are medically eligible will be prescribed bupropion, which they will start two weeks prior to their quit day. Dosage will be 150 mg/daily for days 1-7 and 300 mg/daily (administered in two daily doses) until the 3-month follow-up.
  Other Names: Zyban, Wellbutrin
Drug: nicotine replacement therapy — Participants will be prescribed NRT patch and one nicotine rescue method (e.g., nicotine gum, lozenge, inhaler) for use during the post-quit phase of the study. Participants will be given the choice between nicotine gum, nicotine inhaler, or nicotine nasal spray, and will be instructed to use the rescue method as needed to reduce cigarette cravings
  Other Names: nicotine gum, patch, inhaler, or lozenge
Other: Smoking cessation counseling — Participants will receive four 20-minute smoking cessation counseling sessions and a participant manual. The four sessions are based on standard cognitive-behavioral therapy techniques shown to be efficacious for smoking cessation.
Behavioral: mobile contingency management — Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence. Participants are asked to upload these videos to the study's secured server, and are provided monetary reward for videos that suggest smoking abstinence.
  Other Names: mCM
Other: Stay Quit Coach — Stay Quit Coach is a smart phone application that serves as a source of readily available support and information for adults who are already in treatment to quit smoking and to help them stay quit after treatment. The app guides user in creating tailored plans that include their personal reasons for quitting, interactive tools to help users cope with urges to smoke, motivational messages, support contacts to help users stay smoke free and how to address lapses. Participants assigned to this condition will be asked to use Stay Quit Coach from Session 2 through the 6-month follow-up.
  Other Names: smart phone app
  Arms: QUIT4Ever

SUMMARY:
The primary goal of the study is to evaluate the use of a new smart phone application in preventing relapse to smoking among people with PTSD. The technology intervention will combine a mobile system to reward non-smoking, smoking cessation counseling, smoking cessation medications, and use of the smart phone app. The primary aim is to evaluate how effective this intervention is in preventing smoking relapse compared to another intervention that does not include the app.

DETAILED DESCRIPTION:
The primary goal of the current study will be to evaluate the use of a new smart phone application (app; Stay Quit Coach) in preventing relapse to smoking among individuals with PTSD. The enhanced technology intervention will combine mobile contingency management (mCM), guideline-based smoking cessation counseling, bupropion and nicotine replacement therapy (NRT), and use of the Stay Quit Coach. For this study, we will propose a clinical trial with a two-group design in which 20 smokers with PTSD will be randomized to either:

QUIT4EVER, an intervention that combines guideline-based smoking cessation counseling, bupropion and NRT, mCM and Stay Quit Coach.

COMBINED CONTACT CONTROL (CCC) an intervention that is identical to QUIT4EVER except Stay Quit Coach will not be included. The CCC controls for compensation, monitoring, time and attention effects.

Specific aims are to:

AIM 1: evaluate the efficacy of QUIT4EVER on rates of abstinence from cigarettes (assessed with multiple measures including bioverified abstinence) during short and long term abstinence (measured at 3 and 6 months).

Hypothesis 1: QUIT4EVER will be associated with increased long term abstinence (self-reported and bio-verified prolonged abstinence at the 3 and 6 month follow-up).

AIM 2: assess the impact of QUIT4EVER on counseling treatment completion and medication adherence.

Hypothesis 2. Increased abstinence associated with QUIT4EVER will be partially mediated by increased telephone counseling treatment completion and greater medication adherence.

AIM 3: calculate the relative cost-effectiveness of the QUIT4EVER intervention in quality adjusted life years (QALY).

Hypothesis 3: QUIT4EVER based treatment will result in greater cost-effectiveness compared to the control condition as measured by the incremental cost-effectiveness ratio.

Overall, results of this study could lead to a highly efficient, effective, and easily disseminated treatment method for reducing smoking among smokers with PTSD and other psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Meets criteria for current PTSD;
2. Has current smoking status of at least 10 cigarettes per day (verified with breath carbon monoxide measurement);
3. Has been smoking for at least 1 year;
4. Is aged 18 to 70;
5. Can speak and write current fluent conversation English; and
6. Is willing to make a smoking cessation attempt.

Exclusion Criteria:

1. Is pregnant;
2. Has diagnosis, based on DSM-IV criteria, of schizophrenia, schizophreniform disorder, schizoaffective disorder, current psychotic symptoms, delusional disorder, current (not in remission) substance use disorder, and/or current manic episode;
3. Will not be stable on medications for the study period;
4. Has history of myocardial infarction in past 6 months;
5. Uses any other forms of nicotine such as cigars, pipes, or chewing tobacco with unwillingness to stop use during study period; or
6. Is currently imprisoned.
7. Note: Participants may be excluded or asked to refrain from taking certain study medications if they have a seizure disorder, uncontrolled diabetes, an eating disorder, or current or past cirrhosis or hepatitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
smoking, self-report | 6 months follow-up
  Participants' self-report of smoking in the past seven days will be measured at the end of the treatment intervention, and at 3 and 6-month follow-up contacts.

SECONDARY OUTCOMES:
saliva cotinine | 6 months
  For participants reporting smoking abstinence at 3 and 6-months post treatment follow-ups, we will bio-verify smoking abstinence by collecting saliva samples that will be used to determine salivary cotinine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jean C. Beckham, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Hicks TA Bs, Thomas SP, Wilson SM, Calhoun PS, Kuhn ER, Beckham JC. A Preliminary Investigation of a Relapse Prevention Mobile Application to Maintain Smoking Abstinence Among Individuals With Posttraumatic Stress Disorder. J Dual Diagn. 2017 Jan-Mar;13(1):15-20. doi: 10.1080/15504263.2016.1267828. Epub 2016 Dec 5. PMID 27918881